CLINICAL TRIAL: NCT02438280
Title: Accelerated Tooth Movement With AcceleDent® and Aligners - a Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Greg Huang, Professor, Orthodontics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 49073
Record Dates: First submitted 2015-05-04; First posted 2015-05-08 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-09

CONDITIONS: Tooth Movement; Malocclusion
Keywords: Orthodontic; Orthodontic treatment; Accelerated orthodontics; Vibration
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Vibration (Experimental): Use of Active Vibration (AcceleDent device) 20 minutes each day during treatment with aligners
  Interventions: Device: AcceleDent, Vibrational Device
- Sham Vibration (Active Comparator): Use of Sham Vibration (Sham AcceleDent device) 20 minutes each day during treatment with aligners
  Interventions: Device: AcceleDent, Vibrational Device

INTERVENTIONS:
Device: AcceleDent, Vibrational Device — 20 minutes of vibration each day
  Other Names: AcceleDent Aura

SUMMARY:
The AcceleDent® device has been introduced to the specialty of orthodontics in order to reduce treatment time. The theory behind AcceleDent® is that high frequency vibratory forces (30Hz) delivered to the teeth will stimulate the bone remodeling that is necessary for tooth movement to occur more quickly.

Additionally, one claim of the AcceleDent® product is that it may reduce pain and discomfort during orthodontic treatment.

This study will be a parallel group, triple-blind randomized clinical trial comparing two groups of subjects with 12 participants in each group. Subjects will be randomized to receive one of two vibrational units, which will differ in frequency and/or amplitude of vibration. The subjects will be asked to change their aligners every week instead of every 2 weeks, which is common with Invisalign.

DETAILED DESCRIPTION:
This study will be a parallel group, triple-blind randomized clinical trial comparing two groups of subjects with 12 participants in each group. Subjects will be randomized to receive one of two vibrational units, which will differ in frequency and/or amplitude of vibration. The subjects will be asked to change their aligners every week instead of every 2 weeks, which is common with Invisalign.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malocclusions that require minor or no anterior-posterior or transverse correction in the posterior teeth, and are planned for <= 25 aligners to complete treatment.
2. Treatment must be dual arch in order for patients to qualify for this study.
3. Patients must be 18 years or older

Exclusion Criteria:

1. Patients with systematic diseases or syndromes
2. Patients with a history or current use of Bisphosphonates
3. Patients with current use of nonsteroidal anti-inflammatory drugs (NSAIDs)prostaglandin inhibitors.
4. Patients with generalized moderate to severe periodontitis
5. Patients with active oral hard tissue or soft tissue lesions
6. Patients with chronic oral and maxillofacial conditions such as trigeminal neuralgia, temporomandibular disorder and orofacial pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Huang, Principal Investigator — UW
Locations (3):
- Cohanim Smileworks, Seattle, Washington, United States
- Canada (2):
  - Dr. Sandra Tai, Richmond, British Columbia
  - Dr. Sandra Tai, Vancouver, British Columbia

RESULTS

PARTICIPANT FLOW:
Groups:
- A (Active Device): 20 minutes daily usage in conjunction with orthodontic treatment with clear aligners
  AcceleDent, Vibrational Device: Participants will receive one of two vibrational units
  This groups received Active Devices with frequency of 30Hz ( revealed after study completion )
- B (Control Device): 20 minutes daily usage in conjunction with orthodontic treatment with clear aligners
  AcceleDent, Vibrational Device: Participants will receive one of two vibrational units
  This group received control devices with frequency of 0 Hz ( revealed after study completion )
Period: Overall Study
Arm/Group | A (Active Device) | B (Control Device)
Started | 14 | 13
Completed | 13 | 13
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- A (Active Device); B (Control Device): 20 minutes daily usage in conjunction with orthodontic treatment with clear aligners
  AcceleDent, Vibrational Device: Participants will receive one of two vibrational units
- Total: Total of all reporting groups
Arm/Group | A (Active Device) | B (Control Device) | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 3 | 11
  United States | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Ability to Complete Treatment Aligners in Conjunction With an Active and Placebo Vibration Device (AcceleDent® Aura)
Description: The outcome was the ability to complete the initial set of aligners using either an active vibration device or a placebo vibration device. Regardless of the group assignment, patients were asked to change their aligners each week, and we tracked the percentage that were able to complete their series of aligners.
Time Frame: 6 months
Population: The outcome was the ability to complete the initial set of aligners
Measure: Count of Participants; unit: Participants
Groups:
- A (Active Device): 20 minutes daily usage of an active vibration device
- B (Control Device): 20 minutes daily usage of a placebo vibration device
Arm/Group | A (Active Device) | B (Control Device)
Number analyzed (Participants) | 13 | 13
Participants | 10 | 11

2. Secondary Outcome: Final Alignment Scores of the Upper and Lower Incisors
Description: Final alignment was measured using Little's incisor irregularity index. This index sums the displacement of the contact points of the anterior teeth, to produce a millimetric number. The lower the score, the more perfect the alignment.
Time Frame: 6 months
Population: Final incisor irregularity, measured in millimeters
Measure: Mean (Standard Deviation); unit: Little's irregularity index (mm)
Groups:
- A (Active Device): 20 minutes daily usage of a vibration device
Arm/Group | A (Active Device) | B (Control Device)
Number analyzed (Participants) | 13 | 13
Little's irregularity index (mm) | 2.2 (.92) | 2.1 (.54)

ADVERSE EVENTS:
Time Frame: We collected adverse events data for each patient from the time they began their first aligner until they completed their last aligner, or until they exited the study for some other reason. These periods of time were individual to each patient, as they each had a unique number of aligners, and could have also exited the study if they were not progressing based on the a priori criteria.
Description: We were not expecting any mortality or serious adverse events from the use of the vibrational device. We were monitoring for any other adverse events, like shortening of tooth roots or pain associated with tooth movement. However, we can report that we monitored all patients during the period of the study.
Arm/Group | A (Active Device) | B (Control Device)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
The number of aligners in the upper and lower arches for each patient were made equivalent, in order to end tooth movement at the same time in both arches.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No